CLINICAL TRIAL: NCT03049865
Title: Gait Speed at Discharge as a Marker for Readmission - The GASP Study
Brief Title: Gait Speed at Discharge as a Marker for Readmission
Acronym: GASP
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Holzmann, MD, PhD, Karolinska University Hospital
Other Study IDs: Dnr 2016/2174-31
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: All Disease That May Require Acute Hospitalization Except for Phsychiatric Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The principal aim is to assess if a simple test, the time it takes to walk 10 meters for a patient about to be discharged after a hospital stay for an acute illness, is related to the risk of readmission.

ELIGIBILITY:
Inclusion Criteria:

* >50 years of age Patient discharged to home, or temporary short stay nursing home Expected survival >90 days The ability to read or understand the instructions and to give informed consent.

Exclusion Criteria:

* Planned hospital stay, i.e. the patient was admitted electively The including investigator is directly involved in the care of the patient

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are admitted to hospital from the emergency department are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-09 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Readmission | 30 days

SECONDARY OUTCOMES:
Readmissions | 90,180, 365 days
All-cause mortality | 6, 12, 24, 36, 60 months

IPD SHARING:
Plan to Share IPD: Undecided